CLINICAL TRIAL: NCT05623358
Title: Pharmacist-led Intervention for Optimal Heart Failure Medications: A Pilot Randomized Controlled Trial
Brief Title: PHARM Optimal-HF Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Ricky Turgeon, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H21-01774
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: medication; pharmacist; pharmaceutical care; pharmacotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-led HFrEF medication optimization (Experimental)
  Interventions: Other: Pharmacist-led HFrEF medication optimization; Other: Usual care
- Usual care (Other): Both the intervention group and comparator group will receive usual care by the multidisciplinary HF clinic, including standard-of-care clinical pharmacy services.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pharmacist-led HFrEF medication optimization — In addition to usual care, participants randomized to the intervention arm will receive co-management of medications by a clinical pharmacist with advanced training and expanded scope of practice, with the aim of achieving optimal medical therapy (OMT) for HFrEF as outlined by the 2021 Canadian Cardiovascular Society (CCS) HF guidelines. This will consist of, where possible, the combination of an angiotensin receptor-neprilysin inhibitor (ARNI), evidence-based beta-blocker, mineralocorticoid receptor antagonist (MRA), and sodium-glucose cotransporter 2 inhibitor (SGLT2i) at target doses, along with personalized therapies as outlined in the 2021 CCS HF guidelines, unless the patient is unable to tolerate these agents/doses.
  Arms: Pharmacist-led HFrEF medication optimization
Other: Usual care — Both the intervention group and comparator group will receive usual care by the multidisciplinary HF clinic, including standard-of-care clinical pharmacy services. The standard pathway in the HF clinic consists of an initial consultation with the multidisciplinary team (cardiologist, physician trainees, registered nurse and clinical pharmacist), follow-up visits approximately every 3 months with the nurse and cardiologist until discharge, along with telehealth nurse calls for medication titrations.

SUMMARY:
The goal if this pilot randomized controlled trial is to determine the feasibility of conducting and guide the design of a definitive trial of a pharmacist-led, remotely-administered intervention to optimize medications for heart failure (HF) with reduced ejection fraction (HFrEF) as part of a multidisciplinary HF clinic.

Both the intervention group and comparator group will receive usual care by the multidisciplinary HF clinic, including standard-of-care clinical pharmacy services.

In addition to usual care, participants randomized to the intervention arm will receive co-management of medications by a dedicated study pharmacist with advanced training and expanded scope of practice, with the aim of achieving optimal medical therapy for HFrEF based on the 2021 Canadian Cardiovascular Society HF guidelines. The intervention will consist of 30-minute remote (telephone) encounters with a clinical pharmacist every 1-2 weeks with the aim of initiating or titrating ≥1 medication per encounter using standard protocols, for an intervention duration of up to 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form;
2. Stated willingness to comply with all study procedures and availability for the duration of the study;
3. Age ≥18 years;
4. Clinic diagnosis of HF with New York Heart Association (NYHA) functional class 1 to 3 at time of screening;
5. Left ventricular ejection fraction (LVEF) ≤40% on cardiac imaging performed within 6 months prior to enrolment;
6. Willingness to receive medications for the management of HFrEF;
7. Access to necessary resources for participating (telephone ± computer with internet access).

Exclusion Criteria:

1. Already receiving target doses of sacubitril-valsartan, evidence-based beta-blocker and a mineralocorticoid receptor antagonist at time of screening;
2. Lying/sitting systolic blood pressure <90 mm Hg at time of enrolment;
3. Serum potassium ≥5.5 mmol/L at time of enrolment;
4. ≥2 measurements indicating estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 within 3 months prior to enrolment;
5. Being considered for heart transplant, durable mechanical circulatory support, or intravenous inotropes at time of screening;
6. Requiring diuretic dose greater than furosemide 80 mg equivalents or requiring the addition of a thiazide-like diuretic for more than 3 days at time of screening;
7. Felt by the multidisciplinary HF clinic team to be unsuitable for the trial (e.g. substance abuse and other psychological disorders, significant language barrier).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Baseline
  Composite of:
  1. Proportion eligible at pre-screening ≥50% of all HF clinic patients assessed based on inclusion criteria at pre-screening;
  2. Proportion eligible at screening ≥25% of all patients based on inclusion and exclusion criteria on screening;
  3. Mean recruitment ≥2 participants/week.
Feasibility of achieving rapid optimal medical therapy in intervention arm | month 6
  Feasibility of optimizing HFrEF pharmacotherapy with study intervention, defined as ≥90% attainment of modified OMT score [acceptable] ≥5 at 3 months in intervention arm and ≥80% attainment of modified OMT score 8 [optimal] at 6 months in intervention arm
Feasibility of patient-reported outcome measure (PROM) collection & participant retention | month 12
  Composite of:
  1. Follow-up at 6 months complete in ≥90% at 6 months, ≥80% at 12 months, excluding deaths
  2. ≥90% completion of PROM questionnaires at months 3 and 6, and ≥80% completion at month 12

SECONDARY OUTCOMES:
Optimization of HFrEF medications | month 3
  Modified optimal medical therapy (OMT) score. Range 0 (worst) to 8 (best): suboptimal (0-4), acceptable (5-7), optimal (8).
Optimization of HFrEF medications | month 6
  Modified optimal medical therapy (OMT) score
Optimization of HFrEF medications | month 12
  Modified optimal medical therapy (OMT) score
Medication adherence | month 3
  5-item Medication Adherence Report Scale (MARS-5)
Medication adherence | month 6
  5-item Medication Adherence Report Scale (MARS-5)
Medication adherence | month 12
  5-item Medication Adherence Report Scale (MARS-5)
Medication adverse effects | month 3
  Open-ended question about HF medications
Medication adverse effects | month 6
  Open-ended question about HF medications
Medication adverse effects | month 12
  Open-ended question about HF medications
Quality of life: 12-item Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | month 3
Quality of life: 12-item Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | month 6
Quality of life: 12-item Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | month 12
Treatment burden | month 3
  Treatment Burden Questionnaire (TBQ)
Treatment burden | month 6
  Treatment Burden Questionnaire (TBQ)
Treatment burden | month 12
  Treatment Burden Questionnaire (TBQ)
Treatment satisfaction | month 3
  Treatment Satisfaction with Medicines Questionnaire (SATMED-Q)
Treatment satisfaction | month 6
  Treatment Satisfaction with Medicines Questionnaire (SATMED-Q)
Treatment satisfaction | month 12
  Treatment Satisfaction with Medicines Questionnaire (SATMED-Q)

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Turgeon, BSc(Pharm), ACPR, PharmD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No